CLINICAL TRIAL: NCT05829096
Title: COmbining Brief Interventions for Modifiable Health Behaviours withIN a Physiotherapy Consultation for pEople With a Rotator Cuff Disorder: Development and Testing in a Single-arm Feasibility Study
Brief Title: The COMBINED Study to Integrate Health Behaviour Change for People With a Rotator Cuff Disorder
Acronym: COMBINED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Bury (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor-Investigator, Julie Bury, HEE/NIHR Clinical Doctoral Research Fellow, Manchester Metropolitan University
Organization: Manchester Metropolitan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 51451
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Physiotherapy; Rotator Cuff Syndrome; Rotator Cuff Impingement Syndrome
Keywords: Rotator cuff; Physiotherapy; Shoulder pain; Lifestyle
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Single arm feasibility study
Masking Description: N/A, study does not involve pharmaceutical products or medical devices. There is no randomisation involved in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): This is a single arm interventional study.
  1. A patient-level intervention, which includes:
     * An assessment of existing lifestyle factors (smoking status, physical activity levels, and weight) that may be relevant to shoulder pain;
     * A brief intervention to support health behaviour change with respect to the target behaviours of smoking cessation, increasing physical activity levels and consuming a healthy diet
     * Supporting tools for behaviour change, including an activity workbook for goal-setting and a diary for self-monitoring (attached).
     The intervention is to be delivered by physiotherapists, integrated within a routine consultation for people with a RC disorder.
  2. A clinician-level implementation toolkit to support the delivery of the clinical intervention, which includes a training package and additional resources e.g. scripts to aid conversations with patients.
  Interventions: Other: The COMBINED approach

INTERVENTIONS:
Other: The COMBINED approach — 1. Patient-level intervention:
     * Assessment of existing lifestyle factors (smoking status, physical activity levels, and weight) that may be relevant to shoulder pain;
     * Brief intervention to support health behaviour change: smoking cessation, increasing physical activity levels and consuming a healthy diet
     * Supporting tools for behaviour change, including an activity workbook for goal-setting and a diary for self-monitoring.
  2. Clinician-level implementation toolkit:
     * Training package including a face-to-face workshop, training manual, recorded role play simulations and an online follow-up training session
     * Additional supporting resources; a step-by-step guide to The COMBINED approach, scripts, patient signposting information to support services and a lay summary infographic to explain the links between the health behaviours and RC disorders to patients
     * Audit and feedback via observations of consultations to address any 'drift' from the intervention delivery as intended

SUMMARY:
COMBINED is a pragmatic single-arm feasibility study. The goal of this study is to evaluate the implementation of a physiotherapy-led intervention, The COMBINED approach, to facilitate ongoing refinements, including the strategies for implementation, in readiness for a definitive trial in people with a rotator cuff disorder. The main questions it aims to answer are: 1) What are the key domains of behaviour change influencing the implementation of The COMBINED approach among physiotherapists? 2) Can The COMBINED approach be delivered as intended? 3) Are there any refinements required to the intervention components? 4) What is the patient experience of receiving The COMBINED approach in an NHS setting?

DETAILED DESCRIPTION:
The COMBINED study is looking at how current treatments can be improved for people with shoulder pain, who have been diagnosed with a rotator cuff (RC) disorder. The RC is a group of muscles and tendons which move and stabilise the shoulder joint, and problems with these muscles and tendons can result in pain and difficulty doing everyday tasks.

Current treatments for RC disorders offer only small to moderate benefits and long-term outcomes can be poor. Lifestyle factors, including smoking, being overweight and physical inactivity are associated with the onset and persistence of RC disorders. These factors are linked to modifiable health behaviours that if patients are supported to change, might help improve their shoulder pain. Despite this evidence, physiotherapists do not routinely integrate health behaviour change approaches as part of the management for RC disorders.

The investigators have designed and tested a new complex intervention, The COMBINED approach, that aims to help patients improve their shoulder pain by identifying and assessing the lifestyle factors associated with the onset and persistence of a RC disorder and, where appropriate, the delivery of a brief behaviour change intervention to address these as part of a management plan, supported by a physiotherapist. The investigators have also developed an implementation toolkit to enable and support physiotherapists to effectively deliver this approach in clinical practice. This has been tested and refined in a small usability study, which has led to an optimised version of The COMBINED approach. The investigators would like to find out if this treatment approach can now be delivered within the NHS and to improve this further before testing it in a definitive randomised controlled trial. The overall aim is to provide better care for people with a RC disorder.

This will be a non-randomised feasibility study with qualitative interviews. The study will be conducted in physiotherapy musculoskeletal services across four NHS sites and expected to last 4-6 months. Chartered physiotherapists working at one of the musculoskeletal physiotherapy services, and patients diagnosed with a RC disorder will be eligible to take part.

Physiotherapist participants would be expected to attend a training workshop, deliver the new treatment approach to patients and complete a survey. Patient participants would be asked to attend up to two treatment sessions for their shoulder pain (~60 mins each) with a qualified physiotherapist. During this treatment session they will be asked some questions about their shoulder pain and other things that could be influencing their shoulder pain, such as if they smoke, their weight and how active they are. Where applicable, the physiotherapist may also measure their height and weight during the consultation. The participants will have an examination of their shoulder. Different treatment options will then be discussed. This will be very similar to what participants would expect in a normal physiotherapy appointment. The treatment sessions will be audio-recorded (with consent), for the purpose of checking what information and treatment was delivered by the physiotherapist in the session. The lead researcher may also request (with consent), to observe one of the treatment sessions. The purpose of this is to identify ways to improve how physiotherapists deliver the new treatment approach.

A selection of patients will be asked to take part in an optional short (up to 20 minutes) telephone interview about their views and experience of the treatment session.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the clinician participants are:

* A qualified (HCPC registered) physiotherapist involved in the management of patients with a RC disorder at one of the trial sites;
* Willing to consent to the study procedures, including attending a training workshop, audio-recording of the consultations and audit/feedback on intervention delivery.

The inclusion criteria for patient participants are:

* Adult (aged 18 or over);
* Diagnosed with a RC disorder as per the diagnostic criteria in the British Elbow and Shoulder Society guidelines (Kulkarni et al., 2015), which includes pain mid-range on abduction movement, pain on resisted tests and no loss of external rotation, along with screening of the neck and ruling out other conditions (e.g., instability/frozen shoulder). This will be confirmed by the site Principal Investigators (PI), specialist HCPC registered physiotherapists;
* Able to attend at least one face-to-face physiotherapy consultation. Eligibility will be confirmed via physical examination at this session as per the criteria above;
* Able to give full informed consent;
* Willing to consent to the study procedures, including audio-recording of the consultations.

Exclusion Criteria:

The exclusion criteria for the patient participants are:

* Significant trauma;
* Neurological or inflammatory causes of their shoulder pain;
* Any clinical indications of serious pathology.

We will not exclude anyone based upon protected characteristics for example, age and ethnicity. Anyone referred into the physiotherapy department with a RC disorder will be eligible to take part in the study. Measures in place may include support for the consent process, consultation or patient interviews where required, for example, if verbal translation is needed via a hospital interpreter, personal interpreter or telephone translation service.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
To assess a change in the Determinants of Behavior Questionnaire (DIBQ) | At baseline (0 months) and study completion (expected at 6 months)
  Physiotherapy self-report survey
Fidelity of intervention delivery (self-report checklist by the physiotherapists) will be reported descriptively | 6 months
  What intervention components were delivered by the physiotherapists as intended
Fidelity of intervention delivery (observed through audio-recordings by the research team) will be reported descriptively | 6 months
  What intervention components were delivered by the physiotherapists as intended

SECONDARY OUTCOMES:
Number of patients recruited that have one or more of the identified lifestyle factor will be reported descriptively | 6 months
  Identified lifestyle factors include: Smoker; BMI >25kg/m2; physical activity levels <150/minutes of moderate intensity/week

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bury, Study Chair — Manchester Metropolitan University
Locations (4):
- United Kingdom (4):
  - University Hospitals of Leicester, Leicester, Leicestershire
  - Doncaster and Bassetlaw NHS Foundation Trust, Doncaster, South Yorkshire
  - Calderdale and Huddersfield NHS Foundation Trsut, Halifax, West Yorkshire
  - Airedale Foundation Trust, Keighley, West Yorkshire

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers